CLINICAL TRIAL: NCT02530528
Title: Pilot Trial Assessment of the Antimicrobial Efficacy of Medline 2% CHG Cloth Preoperative Skin Preparation
Brief Title: Pilot Trial of Preoperative Chlorhexidine Gluconate (CHG) Skin Preparation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R13-042
Record Dates: First submitted 2015-08-16; First posted 2015-08-21 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2020-09

CONDITIONS: Surgery
Keywords: Surgical Skin Preparation
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2% CHG 1 min (Experimental): single administration, 1 min application time
  Interventions: Drug: CHG
- 2% CHG 2 min (Experimental): single administration, 2 min application time
  Interventions: Drug: CHG
- 2% CHG 3 min (Experimental): single administration, 3 min application time
  Interventions: Drug: CHG
- Comparator 2% CHG (Active Comparator): Single administration, Marketed CHG
  Interventions: Drug: CHG

INTERVENTIONS:
Drug: CHG — Varied application times
  Other Names: Chlorhexidine Gluconate

SUMMARY:
Pilot study to evaluate and compare activity of investigational preoperative preparation (2% CHG) with comparator (2% CHG).

DETAILED DESCRIPTION:
Evaluate and compare similar preoperative surgical preparations in healthy volunteers. Various application times were evaluated. Efficacy was assess using the Tentative Final Monograph (TFM) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No dermatological conditions

Exclusion Criteria:

* Sensitivity to CHG
* Sensitivity to natural latex rubber or adhesive skin products

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bashir M Hamid, MD, Principal Investigator — Microbac Laboratories

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon achieving sufficient microbial growth prior to product application on either the abdomen, groin or both abdomen and groin regions, sites of the participant were then randomized to receive one or two products for evaluation for up to 4 sites. Differences in the number of participants is based on microbial qualifications.
Pre-assignment Details: Participants were randomized to be treated with at least 2 treatments/Arms (out of 4) at the same time for both groin and abdomen. Numbers represent the total sites tested.
Units Other Than Participants: sites
Groups:
- CHG 1 Min Abdomen; CHG 1 Min Groin: 1 min application time
  CHG: Varied application times
- CHG 2 Min Abdomen; CHG 2 Min Groin: 2 min application time
  CHG: Varied application times
- CHG 3 Min Abdomen; CHG 3 Min Groin: 3 min application time
- Comparator CHG Abdomen; Comparator CHG Groin: Marketed CHG - only applied per products instructions for use
Period: Overall Study
Arm/Group | CHG 1 Min Abdomen | CHG 1 Min Groin | CHG 2 Min Abdomen | CHG 2 Min Groin | CHG 3 Min Abdomen | CHG 3 Min Groin | Comparator CHG Abdomen | Comparator CHG Groin
Started | 13; 13 sites | 13; 13 sites | 14; 14 sites | 14; 14 sites | 13; 13 sites | 13; 13 sites | 14; 14 sites | 14; 14 sites
Completed (27 were treated with both interventions, though interventions differ with application time. 24 subjects completed with passing treatment baseline values.) | 12; 12 sites (13 participants received CHG Cloth) | 12; 12 sites | 12; 12 sites (14 participants received CHG cloth) | 12; 12 sites | 12; 12 sites (13 participants received CHG cloth) | 12; 12 sites | 12; 12 sites (14 participants received comparator CHG.) | 12; 12 sites
Not Completed | 1; 1 sites | 1; 1 sites | 2; 2 sites | 2; 2 sites | 1; 1 sites | 1; 1 sites | 2; 2 sites | 2; 2 sites

BASELINE CHARACTERISTICS:
Population: Number of participants screened
Groups:
- CHG 1, CHG 2, CHG 3, Comparator CHG: Participants could receive up to 2 different treatments at the same time. Treatments included CHG at 1 min, CHG at 2 min, CHG at 3 min or Comparator CHG.
Arm/Group | CHG 1, CHG 2, CHG 3, Comparator CHG
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 32
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 36 [17 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Log Reduction of Bacterial Flora on Abdomen and Groin Sites
Description: Evaluate the Log Reduction of Normal Flora at various sites and timepoints
Time Frame: 10 min, 6 hr and 8 hr
Population: The data represents the number of sites (abdomen/groin) tested.
Measure: Log Mean (Standard Deviation); unit: Log 10 Reduction
Units Other Than Participants: Sites
Groups:
- CHG 1 Min Abdomen; CHG 1 Min Groin: 1 min application time.
- CHG 2 Min Abdomen; CHG 2 Min Groin: 2 min application time.
- CHG 3 Min Abdomen; CHG 3 Min Groin: 3 minute application time
- Comparator CHG Abdomen; Comparator CHG Groin: Comparator CHG solution
Arm/Group | CHG 1 Min Abdomen | CHG 1 Min Groin | CHG 2 Min Abdomen | CHG 2 Min Groin | CHG 3 Min Abdomen | CHG 3 Min Groin | Comparator CHG Abdomen | Comparator CHG Groin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Number analyzed (Sites) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Log 10 Reduction
  10 min | 2.6 (0.65) | 3.4 (0.85) | 2.7 (0.60) | 4.2 (1.3) | 2.8 (0.46) | 4.3 (1.2) | 2.6 (0.71) | 3.1 (0.79)
  6 hour | 2.0 (0.86) | 2.7 (0.67) | 2.4 (0.80) | 2.9 (1.13) | 2.4 (0.81) | 3.5 (0.95) | 1.9 (0.64) | 2.7 (1.0)
  8 hour | 1.9 (0.76) | 2.9 (0.38) | 2.4 (1.0) | 3.05 (0.83) | 1.9 (0.67) | 3.2 (0.8) | 1.6 (0.94) | 2.5 (0.94)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline out to 8 hours.
Description: Participants received up to 2 products at the same time.
Groups:
- CHG 1 Min: 1 min application time
- CHG 2 Min: 2 min application time
- CHG 3 Min: 3 minute application time
- Comparator CHG: Instructions for use
Arm/Group | CHG 1 Min | CHG 2 Min | CHG 3 Min | Comparator CHG
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data remains confidential